CLINICAL TRIAL: NCT07351916
Title: Remission in Adults With Mild-to-moderate Asthma in Thailand
Status: Not yet recruiting | Type: Observational
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Narongkorn Saiphoklang, MD, Associate Professsor, Thammasat University
Other Study IDs: MTU-EC-IM-0-282/68
Record Dates: First submitted 2026-01-10; First posted 2026-01-20 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Asthma; Mild-to-moderate Asthma; Asthma Control Level
Keywords: asthma; asthma control; mild-to-moderate asthma; Thailand; remission; FeNO; blood eosinophil count
MeSH Terms: conditions — Asthma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mild-to-moderate asthma: Patients aged 18 years or older with mild-to-moderate asthma. Mild asthma refers to asthma patients who experience symptoms <3 times per week, have preserved lung function (FEV₁ or PEF >80% of predicted), and whose symptoms can be adequately controlled with low-dose inhaled corticosteroids (low-dose ICS) alone, without the need for long-acting bronchodilators or other controller medications.
  Moderate asthma refers to asthma patients who have symptoms >4-5 days per week or experience nocturnal asthma symptoms >1 per week, and who require treatment with medium-dose inhaled corticosteroids (medium-dose ICS) or low-dose ICS in combination with a long-acting β₂-agonist (low-dose ICS/LABA) to achieve symptom control and prevent exacerbations.
  Interventions: Other: Global Initiative for Asthma (GINA) and Asthma Control Test (ACT) questionnaires; Other: Spirometry; Other: Fractional exhaled nitric oxide (FeNO) test; Other: Blood eosinophil count (BEC)

INTERVENTIONS:
Other: Global Initiative for Asthma (GINA) and Asthma Control Test (ACT) questionnaires — GINA and ACT are questionnaires used to assess the level of asthma control.
Other: Spirometry — Spirometry is a tool used to assess pulmonary function.
Other: Fractional exhaled nitric oxide (FeNO) test — FeNO is a tool used to assess eosinophilic airway inflammation and asthma remission.
Other: Blood eosinophil count (BEC) — BEC is a tool used to assess eosinophilic inflammation and asthma remission.

SUMMARY:
The goal of this observational study is to determine the prevalence of remission among adults with mild-to-moderate asthma, as well as the factors associated with remission in Thailand.

The main question the study aims to answer is:

What is the prevalence of remission among adults with severe asthma in Thailand? Participants will complete a questionnaire on asthma symptoms and undergo pulmonary function testing and a blood test once.

DETAILED DESCRIPTION:
This study is a cross-sectional study. Thai patients aged 18 years or older with mild-to-moderate asthma are included in the study. Participants will complete two questionnaires about asthma control: the Global Initiative for Asthma (GINA) and the Asthma Control Test (ACT), and will perform spirometry, a fractional exhaled nitric oxide (FeNO) test, and blood eosinophil counts (BEC).

GINA and ACT are questionnaires used to assess the level of asthma control.

ELIGIBILITY:
Inclusion Criteria:

* mild-to-moderate asthma
* age 18 years or older

Exclusion Criteria:

* inability to perform spirometry or fractional exhaled nitric oxide (FeNO) test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thai patients aged 18 years or older with mild-to-moderate asthma are included in the study
Sampling Method: Non-Probability Sample
Enrollment: 289 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence rate of mild-to-moderate asthma remission | An average of 1 year
  Prevalence rate of mild-to-moderate asthma remission (%)

SECONDARY OUTCOMES:
Asthma control in patients with mild-to-moderate asthma | At baseline and at 12 months
  Rate of patients with well-controlled asthma. Well-controlled asthma is defined as an Asthma Control Test (ACT) score of 20 or higher.
Airway obstruction in patients with mild-to-moderate asthma | At baseline and at 12 months
  Airway obstruction is assessed using FEV1/FVC ratio on spirometry.
Severity of aiway obstruction in patients with mild-to-moderate asthma | At baseline and at 12 months
  The severity of aiway obstruction is assessed using FEV1 % predicted on spirometry.
Eosinophil airway inflammation in patients with mild-to-moderate asthma | At baseline and at 12 months
  Eosinophil airway inflammation is assessed using blood eosinophil count (cells/µL).
Type 2 airway inflammation in patients with mild-to-moderate asthma | At baseline and at 12 months
  Type 2 airway inflammation is assessed using fractional exhaled nitric oxide (FeNO, ppb).

CONTACTS AND LOCATIONS:
Overall Officials: Narongkorn Saiphoklang, MD, Principal Investigator — Thammasat University Faculty of Medicine
Locations (1):
- Faculty of Medicine, Thammasat University, Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: Yes
IPD and documents will be available for sharing immediately after publication for a period of 2 years.
Supporting Information: Study Protocol, SAP
Time Frame: IPD and documents will be available for sharing immediately after publication for a period of 2 years.

REFERENCES:
- [Result] Ishizuka M, Sugimoto N, Kobayashi K, Takeshita Y, Imoto S, Koizumi Y, Togashi Y, Tanaka Y, Nagata M, Hattori S, Uehara Y, Suzuki Y, Toyota H, Ishii S, Nagase H. Clinical remission of mild-to-moderate asthma: Rates, contributing factors, and stability. J Allergy Clin Immunol Glob. 2025 Jan 30;4(2):100431. doi: 10.1016/j.jacig.2025.100431. eCollection 2025 May. PMID 40091885
- [Result] Holm M, Omenaas E, Gislason T, Svanes C, Jogi R, Norrman E, Janson C, Toren K; RHINE Study Group. Remission of asthma: a prospective longitudinal study from northern Europe (RHINE study). Eur Respir J. 2007 Jul;30(1):62-5. doi: 10.1183/09031936.00121705. Epub 2007 Mar 14. PMID 17360725
- [Result] Tupper OD, Hakansson KEJ, Ulrik CS. Remission and Changes in Severity Over 30 Years in an Adult Asthma Cohort. J Allergy Clin Immunol Pract. 2021 Apr;9(4):1595-1603.e5. doi: 10.1016/j.jaip.2020.11.013. Epub 2020 Nov 19. PMID 33220516
- [Result] Chiewchalermsri C, Kanjanawasee D, Saiphoklang N, Chirakalwasan N, Sriprasart T, Senavonge A, Sanguanwong N, Kamalaporn H, Athipongarporn A, Hachai S, Boonsawat W, Brannan JD, Song WJ, Ruxrungtham K, Poachanukoon O. Asthma remission: A path to cure? Asian Pac J Allergy Immunol. 2025 Jun;43(2):135-150. doi: 10.12932/AP-240525-2082. PMID 40652405